CLINICAL TRIAL: NCT06276582
Title: Screening for Neonatal Jaundice With a Mobile Health Device: a Validation Study in Oaxaca, Mexico.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Picterus AS (Industry); Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 519379-2
Record Dates: First submitted 2024-02-05; First posted 2024-02-26 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Jaundice, Neonatal
Keywords: Neonatal jaundice; Screening; mobile health; low resource settings
MeSH Terms: conditions — Jaundice, Neonatal | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening for neonatal jaundice with a mobile health device (Experimental): Neonatal jaundice will be screened using the app Picterus JP and the results will be compared to the total serum bilirubin level from a blood test.
  Interventions: Device: Screening for neonatal jaundice with a mobile health device

INTERVENTIONS:
Device: Screening for neonatal jaundice with a mobile health device — Picterus Jaundice Pro will be used to screen for neonatal jaundice by taking 6 photos of the newborns skin, where the Picterus calibration card is place.

SUMMARY:
The performance and accuracy of the smartphone application (app) Picterus Jaundice Pro (PicterusJP) will be validated by a cross-sectional study conducted in low resource settings in Mexico. Physics-based and machine learning-based models will be used to analyze the images obtained with the app and its performance will be compared.

DETAILED DESCRIPTION:
A cross-sectional prospective study is taken place at Hospital General de Zona 1 in the city of Oaxaca, Mexico.

Participants are recruited from the maternity ward and emergency room and data collection is conducted by one experienced pediatrician and one paediatrics' resident. After informed consent is obtained, background data including time and date or birth, birth weight, gestational age, parent's skin type according to Fitzpatrick scale and newborn's skin color according to Neomar's scale is being collected. Visual assessment is performed by the researchers using Kramer's scale. To obtain the bilirubin measurements with the smartphone app Picterus Jaundice Pro (Picterus JP), the calibration card is placed on the newborn's chest and a set of six images, 3 with and 3 without flash, are captured. The smartphones used to capture the images are Samsung A23, iPhone 11 and iPhone 15 Pro.

Total serum bilirubin (TSB) levels are measured with a blood sample obtained within one hour of capturing the images and analyzed at the hospital laboratory facilities.

Demographic and clinical characteristics will be analyzed by descriptive statistic.

Bilirubin measurements correlation between Picterus JP using both models and TSB will be determined by Pearson's correlation coefficient. Systematic over or underestimation of bilirubin levels will be evaluated using Bland-Altman plots. Accuracy measurements will be determined using receiver operating characteristics (ROC) and area under the curve (AUC) analysis. To compare the correlations from both models, Fisher's r to z transformation approach will be applied

ELIGIBILITY:
Inclusion Criteria:

* gestational age of 37 weeks or more
* birth weight of 2500 g and above
* newborns in whom a blood test had been ordered for any reason, irrespective of the study

Exclusion Criteria:

* newborns with congenital diseases
* newborns transferred to pediatric wards for reasons unrelated to neonatal jaundice
* newborns who had undergone phototherapy

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 177 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-06-08 (Actual); Study Completion 2024-06-08 (Actual)

PRIMARY OUTCOMES:
Enable high qualitative estimation of bilirubin levels in the blood of Mexican newborns using Picterus JP | 16 months
  Evaluate the smartphone-based screening tool Picterus for neonatal jaundice in Mexican newborns.

SECONDARY OUTCOMES:
Correlation between bilirubin measurements with Picterus JP and total serum bilirubin | 2 hours
  Pearson correlation coefficient

OTHER OUTCOMES:
Accuracy of Picterus JP to screen for neonatal jaundice | 16 months
  Sensitivity, specificity, positive and negative predictive values

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General de Zona 1, Oaxaca City, Mexico

REFERENCES:
- [Derived] Jimenez-Diaz G, Gierman LM, Keitsch M, Elizarraras-Rivas J, Silva-Mendez RM, Infanti JJ, Marcuzzi A. Validation of a Mobile Health Device for Neonatal Jaundice Screening: A Cross-Sectional Study in a Resource-Limited Setting in Mexico. Sage Open Pediatr. 2025 Apr 22;12:30502225251320544. doi: 10.1177/30502225251320544. eCollection 2025 Jan-Dec. PMID 40612198